CLINICAL TRIAL: NCT04011423
Title: Effects of Combined Whole Body Vibration and Unstable Shoes on Balance in Healthy Young People: A Preliminary Randomized Controlled Trial
Brief Title: Whole Body Vibration and Unstable Shoes on Balance in Healthy Young People
Acronym: WBV-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-24
Record Dates: First submitted 2019-07-05; First posted 2019-07-08 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Balance
Keywords: Unstable Shoes; Whole Body Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unstable shoes (Experimental): Wearing unstable shoes during the whole-body vibration training
  Interventions: Other: Unstable shoes plus Whole-body vibration
- Stable shoes (Active Comparator): Wearing stable shoes during the whole-body vibration training
  Interventions: Other: Stable shoes plus Whole-body vibration

INTERVENTIONS:
Other: Unstable shoes plus Whole-body vibration — Wearing unstable shoes during the whole-body vibration training
  Arms: Unstable shoes
Other: Stable shoes plus Whole-body vibration — Wearing stable shoes during the whole-body vibration training
  Arms: Stable shoes

SUMMARY:
Aim: To compare the effect of different type of shoes (unstable or stable) combined with a whole body vibration training on balance.

Design: Randomized controlled trial.

Setting: Laboratory of biomechanics.

Population: Healthy young people.

DETAILED DESCRIPTION:
Background: The use of whole body vibration to train strength and balance has increased in the last years. Last studies have shown that adding an unstable device increased electromyographic activity of the lower limb and the trunk muscles. However, no studies have investigated the effects of wearing unstable shoes during a whole-body vibration training on balance in healthy young people.

Aim: To compare the effects of different type of shoes (unstable [Intervention group] or stable [Control group]) combined with a 12-weeks whole body vibration training on balance.

Setting: Laboratory of biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 35.

Exclusion Criteria:

* Cardiovascular disease, incapacity to practice a physical activity, musculoskeletal pathologies, neurologic diseases, previous experience with unstable shoes, previous experience with whole-body vibration.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Balance | 4 weeks
  Velocity of the center of pressure assessed with a foot pressure sensitive walkway

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Salvador-Coloma P, Arguisuelas MD, Domenech-Fernandez J, Sanchez-Zuriaga D, Amer-Cuenca JJ, Martinez-Gramage J, Montanez-Aguilera FJ, Lison JF. Effects of unstable shoes on trunk muscle activity in patients with chronic low back pain. Gait Posture. 2018 Jul;64:165-168. doi: 10.1016/j.gaitpost.2018.06.025. Epub 2018 Jun 11. PMID 29909231
- [Result] Lison JF, Ortega-Santana B, Anton-Nogues A, Gonzalez-Requena P, Vera-Hervas C, Domenech-Fernandez J, Sanchez-Zuriaga D, Salvador-Coloma P. Effects and underlying mechanisms of unstable shoes on chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 May;32(5):654-662. doi: 10.1177/0269215517753972. Epub 2018 Jan 14. PMID 29333872